CLINICAL TRIAL: NCT06334809
Title: Identification of Genomic Screening Pathways in Cancer Patients With DNA Repair Alterations
Brief Title: INSIDE: Identification of Genomic Screening Pathways in Cancer Patients With DNA Repair Alterations
Acronym: INSIDE
Status: Recruiting | Type: Observational
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: 028FPO22
Record Dates: First submitted 2024-02-16; First posted 2024-03-28 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; mHSPC; castration-resistant; PARP inhibitory; mCRPC
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — will be collected: one test tube of ctDNA before the radical biomedical treatment, one will be collected after 6 and 12 months and at the time of progression. A representative sample of archival tumor tissue from diagnostic biopsy/prostatectomy and a biopsy of the metastasis will also be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort A:patients with high risk localized prostate cancer: Cohort A:150 patients with high risk localized prostate cancer (defined as >cT3 or PSA > 20 ng/mL or presence of ECE or SVIat mpMRI), with tissue available from diagnostic biopsy/prostatectomy undergoing or who underwent curative treatment (prostatectomy/radical radiotherapy) but have not started a FU pathway.
  Patients within Cohort A will be followed up with PSA every 3 months for 3 years and early scans. They will also receive a blood sample for ctDNA/CTC before (when feasible) and after radical treatment, 6 months and 12 months (if not progressed), at time of PSA or radiological progression
- Cohort B: patients with de novo metastatic hormone sensitive prostate cancer (mHSPC): Cohort B: 100 patients with de novo metastatic hormone sensitive prostate cancer (mHSPC) with tissue available from diagnostic biopsy of the primary and when possiblepossible, from a metastatic site. Patients must either have not started a standard treatment or have started for not longer than 3 months;Patients within Cohort B will be followed up with PSA and scans every 3 months. They will also receive a blood sample before (when feasible) or after the start of systemic treatment, 6 months and 12 months (if not progressed), at time of PSA or radiological progression
- Cohort C:Patients with metastatic castration resistant prostate cancer (mCRPC) progressing: Cohort C:100-150 patients with metastatic castration resistant prostate cancer tissue (mCRPC) progressing on a standard treatment with available from biopsy of a metastatic site, and when possiblepossible, from the primary.Patients within Cohort C will be followed up with PSA monthly and scans every 3 month. They will also receive a blood sample for ctDNA/CTC before (when feasible) or after the start of systemic treatment, 6 months and 12 months (if not progressed), at time of PSA or radiological progression.

SUMMARY:
400 patients will be enrolled and divided into 3 cohorts: Cohort A: patients with high risk localized prostate cancer (PC) defined as >cT3 or PSA > 20 ng/mL or presence of ECE or SVI at mpMRI;

Cohort B: patients with de novo metastatic hormone sensitive prostate cancer (mHSPC);

Cohort C: patients with metastatic castration resistant prostate cancer (mCRPC) progressing on a standard treatment.

DETAILED DESCRIPTION:
In this study 150 patients will be enrolled in cohort A, 100 patients in cohort B and 100-150 patients in Cohort C.

Considering the known frequency of DDR and MMR germline/somatic alterations, it is expected to see:

* 15-23 patients with germline/somatic DDR defects and 5-7 MMR alterations in cohort A;
* 20-25 patients with germline/somatic DDR defects and 5-7 MMR alterations in cohort B;
* 25-35 patients with germline/somatic DDR defects and 7-10 MMR alterations in cohort C.

Patients within Cohort A will be followed up with PSA every 3 months for 3 years and early scans. They will also receive a blood sample for ctDNA/CTC before (when feasible) and after radical treatment, 6 months and 12 months (if not progressed), at time of PSA or radiological progression;

Patients within Cohort B will be followed up with PSA and scans every 3 months. They will also receive a blood sample before (when feasible) or after the start of systemic treatment, 6 months and 12 months (if not progressed), at time of PSA or radiological progression.

Patients within Cohort C will be followed up with PSA monthly and scans every 3 month. They will also receive a blood sample for ctDNA/CTC before (when feasible) or after the start of systemic treatment, 6 months and 12 months (if not progressed), at time of PSA or radiological progression.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of prostate cancer as indicated below:

Cohort A: patients with high risk localized prostate cancer (defined as >cT3 or PSA > 20 ng/mL or presence of ECE or SVIat mpMRI), with tissue available from diagnostic biopsy/ prostatectomy undergoing or who underwent curative treatment (prostatectomy/ radical radiotherapy) but have not started a FU pathway.

Cohort B: patients with de novo metastatic hormone sensitive prostate cancer (mHSPC) with tissue available from diagnostic biopsy of the primary and when possiblepossible, from a metastatic site. Patients must either have not started a standard treatment or have started for not longer than 3 months.

Cohort C: patients with metastatic castration resistant prostate cancer tissue (mCRPC) progressing on a standard treatment with available from biopsy of a metastatic site, and when possiblepossible, from the primary.

* Ability to understand and consent to informed consent;
* Patient must be compliant with receiving a biopsy of the metastatic site (cohort C) and with FU assessments schedule

Exclusion Criteria:

• Patients not willing to comply with study's procedures or fulfilling the inclusion criteria.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort A: patients with high risk localized prostate cancer (PC) defined as >cT3 or PSA > 20 ng/mL or presence of ECE or SVI at mpMRI; Cohort B: patients with de novo metastatic hormone sensitive prostate cancer (mHSPC); Cohort C: patients with metastatic castration resistant prostate cancer (mCRPC) progressing on a standard treatment.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number, type and frequency of DDR and MMR germline/somatic alterations | 24 months
  Evaluation of the frequency, number and type of DDR and MMR germline/somatic alterations in the study population
Changes in PSA levels in the 3 cohorts | 36 months
  Evaluation of PSA levels (baseline versus follow-up) in the 3 cohorts compared with radiological assessment

SECONDARY OUTCOMES:
Number of patient-derived preclinical models | 36 months
  Number of patient-derived preclinical models (primary 2D cell lines, organoids or PDXs)

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Rescigno, MD, Principal Investigator — Fondazione del Piemonte per l'Oncologia-IRCCS Candiolo; Sabrina Arena, PhD, Principal Investigator — Fondazione del Piemonte per l'Oncologia-IRCCS Candiolo
Locations (2):
- Italy (2):
  - Fondazione del Piemonte per l'Oncologia-IRCCS Candiolo, Candiolo, Turin
  - AOU San Luigi Gonzaga, Orbassano, Turin